CLINICAL TRIAL: NCT00308568
Title: Randomized Controlled Trial of a Mailed Brochure to Increase Adherence to Referrals for Screening Colonoscopy
Brief Title: RCT of Mailed Brochure to Boost Adherence to Screening Colonoscopy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Colorado, Denver (Other)
Collaborators: The Henry J. Kaiser Family Foundation (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 05-0038; MRSG-06-081-01-CPPB-01 (Other)
Record Dates: First submitted 2006-03-27; First posted 2006-03-29 (Estimated); Last update posted 2017-05-04 (Actual); Status verified 2017-05

CONDITIONS: Colonoscopy; Mass Screening
Keywords: screening colonoscopy; adherence

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: Mailed educational brochure

SUMMARY:
The purpose of this study is to evaluate the effect of a mailed educational brochure on adherence to referral for screening colonoscopy. The comparison (or control) group receives no mailer, which is usual care.

ELIGIBILITY:
Inclusion Criteria:

Referrals for screening colonoscopy; Asymptomatic; age>=50

Exclusion Criteria:

Referrals for diagnostic colonoscopy

Min Age: 50 Years | Sex: All
Age Groups: Adult, Older Adult
Enrollment: 628
Dates: Start 2006-02; Primary Completion 2006-03 (Actual); Study Completion 2006-03 (Actual)

PRIMARY OUTCOMES:
Rate of adherence to screening colonoscopy referral within at least three months of receipt of referral.

CONTACTS AND LOCATIONS:
Overall Officials: Thomas D. Denberg, MD, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- University of Colorado at Denver and Health Sciences Center, Denver, Colorado, United States

IPD SHARING:
Plan to Share IPD: No
only through publication in journals, this is not an applicable clinical trial